CLINICAL TRIAL: NCT03243903
Title: The Safety and Efficacy of QS-M Needle -Free Injector Versus Needle-insulin Pen as a Drug Carrier for Controlling the Blood Glucose in T2DM：a Randomized, Parallel Controlled, Open-label, Multicenter Trial
Brief Title: Comparison of Safety and Efficacy of QS-M Needle- Free Injector and Insulin Pen in Controlling T2DM Patient's Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing QS Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSE01
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Diabetes
Keywords: T2DM; QS-M needle free injector; insulin pen; effective; safety
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- needle-free insulin injector (Experimental): Using QS-M insulin-free injector as insulin carrier to control blood glucose of T2DM and insulin dose is prescribed.
  Interventions: Device: QS-M insulin-free injector
- conventional insulin pen (Active Comparator): Using conventional insulin pen as insulin carrier to control blood glucose of T2DM and insulin dose is prescribed.
  Interventions: Device: conventional insulin pen

INTERVENTIONS:
Device: QS-M insulin-free injector — Using QS-M insulin-free injector as insulin carrier to control blood glucose of T2DM and insulin dose is prescribed.
  Arms: needle-free insulin injector
Device: conventional insulin pen — Using conventional insulin pen as insulin carrier to control blood glucose of T2DM and insulin dose is prescribed.
  Arms: conventional insulin pen

SUMMARY:
In this study, QS-M needle-free injector and needle-insulin pen were used as a drug carrier to control blood glucose in type 2 diabetic patients（T2DM）.The efficacy and safety of QS-M needle-free injector and needle-insulin pen were evaluated and compared.This is a needle-insulin pen as control group, using a prospective, multicenter, randomized, open, parallel grouping study.

DETAILED DESCRIPTION:
The research purpose is to evaluate the efficacy and safety of QS-M needle-free injector as a drug carrier in the control of blood glucose in patients with type 2 diabetes mellitus by non-inferiority study，using needle-insulin pen as the comparison. This is a prospective, multicenter, randomized, open and parallel grouping study. QS-M needle-free injector produced by Beijing QS medical technology co., Ltd.is used as the insulin carrier in the experimental group. While needle-insulin pen is used as the insulin carrier in the control group. In this study, the investigators investigated whether the changes of glycosylated hemoglobin (HbA1c) at the 16th week in the experimental group respected to the baseline is non-inferiority compared with that in control group. A total of 427 patients with T2DM were enrolled in a prospective, multicenter,randomized, open-label study, and were randomly assigned 1:1 to receive 16 weeks' treatment with basal insulin or premixed insulin administered either by a needle-free insulin injector (NFII)or insulin treatment via a conventional insulin pen (CIP)

Patients in both groups entered a 2-week screening period after providing their written informed consent. A run-in period from week 1 to the end of week 4 was implemented to allow treatment adjustment. Assessment visits occurred at screening (week -2), baseline, and week 1, 2, 4, 6, 8, 12 and 16.After the 4-week run-in phase, the patients entered a 12-week treatment observation period. All patients were unable to change the type of insulin and the number of injections during the study period. In this study, the treatment regimen was adjusted according to the results of the determination of prescription blood glucose. According to clinical experience, the adjustment of blood glucose fluctuations in the possibility of a larger, so the study of the adjustment phase follow-up frequency is greater than the treatment period.

Explanation of Visits and Timing of Assessments:

Baseline assessment was performed for all subjects during the screening period. On the first day of treatment, the first week after treatment (± 2 days), the second week (± 2 days), the 4th week (± 5 days), the 6th week (± 5 days), the 8th week (± 5 days),the 12th week (± 5 days), the 16th week (± 5 days) for visit.The 3th week (± 2 days), the 5th week (± 5 days), the 7th week (± 5 days), the 10th week (± 5 days), the 14th week (± 5 days), for telephone interviews.

ELIGIBILITY:
Inclusion Criteria:

1. have been diagnosed with type 2 diabetes; (A) have been treated with insulin (premixed or basal) subcutaneous injection therapy (without limitation or combined oral hypoglycemic agents); (B) the subjects with poor blood sugar control is taking oral hypoglycemic agents or living interventions need Initiating insulin therapy (see Appendix 1 for initiating treatment regimens);
2. adults aged 18-75 years, women of childbearing age need to take adequate contraceptive measures to reduce the pregnancy risk to the minimum;
3. injection of insulin and / or oral hypoglycemic agents ≥ 3 months before enroll the study, the insulin dose adjustment ≤ 10% within 1 month before enrolling (adjustment = (the maximum dose within a month - the minimum dose) / Final dose (dose of the day before the visit) × 100%);
4. have a HbAlc value (detected by NGSP approved method) between 7.5-11% ;
5. BMI ≤ 32kg / m2, the body weight remained relatively stable, body weight change of no more than 10% at least 3 months before screening,
6. Male subjects hemoglobin≥12g/dl (≥ 120g / L), female subjects hemoglobin ≥ 11g / dl (≥ 110g / L);
7. serum creatinine <1.5 mg / dL for male subjects, serum creatinine <1.4 mg / dL for female subjects;
8. have not participated in other clinical studies related diabetes treatment within 3 months ;
9. be volunteered to participate in this clinical study and signed informed consent.

Exclusion Criteria:

1. the persons who attend or perform this study;
2. women in pregnancy or lactation;
3. have frequent severe hypoglycaemia in one month; have blood glucose control adverse events like diabetic ketoacidosis or hyperosmotic diabetic coma within half a year;
4. have severe cardiovascular events in the past 6 months, such as myocardial infarction, acute coronary syndrome, cerebral infarction, cardiovascular and cerebrovascular surgery;
5. have used hormones or immunosuppressive agents, or have immunologic deficiency disease;
6. have end-stage renal disease, and are receiving dialysis treatment;
7. have of history of cancer within 5 years;
8. have history of severe mental instability;
9. have long-term alcohol abuse or drug abuse history;
10. have Skin lesions in the insulin injection site;
11. have history of anemia caused by hemoglobinopathy (such as sickle cell red blood cell anemia, thalassemia, sideroblastic anemia) or any other course;
12. have critically ill, or life expectancy is less than one year;
13. difficult to evaluate the effectiveness and safety of the device intervention;
14. have a clear infection history within a month, such as pneumonia;
15. have active liver disease (AST> 3 times of normal upper limit or ALT> 3 times of normal upper limit);
16. have history of acute pancreatitis within a month;
17. have history of insulin allergy;
18. have been expected to have poor compliance and can not be treated according to the research protocol;
19. other cases that investigators believe that the subject may fail to complete the study or may have a significant impact.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
glycosylated hemoglobin (HbA1c) | 16weeks
  The changes in glycosylated hemoglobin (HbA1c) value between the 16th week of treatment and the start of the adjustment period (using NGSP approved detection method to detect the glycosylated hemoglobin values) .

SECONDARY OUTCOMES:
Self-monitoring of blood glucose(SMBG) | 16 weeks
  SMBG blood glucose value (on the first day and two days before the 1st, 2nd, 4th, 6th, 8th, 12th, 16th weeks interview, test the values before and 2 hours after the three meals and before sleeping).

OTHER OUTCOMES:
The rate of glycosylated hemoglobin | 16 weeks
  The rate of glycosylated hemoglobin (according to the percentage of HbA1c <7.0% of the total number of subjetcs at 16th weeks).
SF-36 | 16 weeks
  Quality of Life Questionnaire (SF-36) (the changes comparison about SF-36 quality of life score between 16th weeks of subjects and baseline.
Insulin dose | 16 weeks
  Insulin dose (the actual total dose of injected insulin of the first day and the day before the 1st,2nd,4th,6th,8th,12th,16th weeks' interview).
Insulin treatment compliance | 16 weeks
  Insulin treatment compliance (recording whether the subjects obey the program to inject insulin at the specified time point in the 1st, 2nd, 4th, 6th, 8th, 12th, 16th weeks).
Subject Satisfaction | 16weeks
  Subject Satisfaction ( the 16th Week overall satisfaction for the use of injectable equipment). At the end of the trial (16th week),recording and comparing the experimental group / control subjects the overall satisfaction of the injector used in the trial. According to the subjective satisfaction to scoring, the satisfaction score form 0 to 10. With the minimum score 0 for the least satisfied and the maximum score 10 for the most satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Li Nong, Principal Investigator — Peking University People 's Hospital
Locations (1):
- Peking University People 's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ji L, Gao L, Chen L, Wang Y, Ma Z, Ran X, Sun Z, Xu X, Wang G, Guo L, Shan Z. Insulin delivery with a needle-free insulin injector versus a conventional insulin pen in Chinese patients with type 2 diabetes mellitus: A 16-week, multicenter, randomized clinical trial (the FREE study). EClinicalMedicine. 2020 Jun 4;23:100368. doi: 10.1016/j.eclinm.2020.100368. eCollection 2020 Jun. PMID 32529176
- [Derived] Ji L, Chen L, Wang Y, Ma Z, Ran X, Sun Z, Xu X, Wang G, Guo L, Shan Z. Study Protocol for a Prospective, Multicenter, Randomized, Open-Label, Parallel-Group Clinical Trial Comparing the Efficacy and Safety of a Needle-Free Insulin Injector and a Conventional Insulin Pen in Controlling Blood Glucose Concentrations in Chinese Patients with Type 2 Diabetes Mellitus (The FREE Study). Adv Ther. 2019 Jun;36(6):1485-1496. doi: 10.1007/s12325-019-00951-4. Epub 2019 Apr 19. PMID 31004325